CLINICAL TRIAL: NCT01333709
Title: A Randomized Multicenter Phase 2 Study: a Tailored Strategy for Locally Advanced Rectal Carcinoma
Brief Title: Multicenter Phase 2 Trial: a Tailored Strategy for Locally Advanced Rectal Carcinoma
Acronym: GRECCAR4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRECCAR 4; 2010-023546-73 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Locally Advanced Malignant Neoplasm; Rectal Carcinoma
Keywords: locally advanced rectal carcinoma; Tailored treatment strategy; MRI volumetry; Early tumor response
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A: immediate rectal surgery (Experimental): "Very good" responder patients will be randomly assigned to proctectomy within 2-4 weeks after the end of the induction chemotherapy.
  Interventions: Drug: Induction trichemotherapy - FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Procedure: Radical proctectomy with total mesorectal excision
- Arm B: RCT Cap 50 and then rectal surgery (Other): "Very good" responder patients will be randomly assigned to receive chemoradiotherapy combining the administration of oral capecitabine (1600 mg/m2/day, BID) and radiotherapy at a total dose of 50 grays (2Gy/day, 5 days a week, 5 weeks, boost 6 Gy).
  Interventions: Drug: Induction trichemotherapy - FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Radiation: Radiochemotherapy Cap 50; Procedure: Radical proctectomy with total mesorectal excision
- Arm C: RCT Cap 50 and then rectal surgery (Other): "Good or poor" responder patients will be randomly assigned to receive chemoradiotherapy combining the administration of oral capecitabine (1600 mg/m2/day, BID) and radiotherapy at a total dose of 50 grays (2Gy/day, 5 days a week, 5 weeks, boost 6 Gy).
  Interventions: Drug: Induction trichemotherapy - FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Radiation: Radiochemotherapy Cap 50; Procedure: Radical proctectomy with total mesorectal excision
- Bras D: RCT Cap 60 and then rectal surgery (Experimental): "Good or poor" responder patients will be randomly assigned to receive chemoradiotherapy combining the administration of oral capecitabine (1600 mg/m2/day, BID) and radiotherapy at a total dose of 60 grays (2Gy/day, 5 days a week, 6 weeks, boost 14 Gy).
  Interventions: Drug: Induction trichemotherapy - FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Radiation: Radiochemotherapy Cap 60; Procedure: Radical proctectomy with total mesorectal excision

INTERVENTIONS:
Drug: Induction trichemotherapy - FOLFIRINOX regimen — A short (4 cycles) and intensive trichemotherapy combinig irinotecan 180 mg/m2, oxaliplatin 85 mg/m2, elvorin 200 mg/m2, 5-Fu (bolus 400 mg/m2, followed by a 46-hour continuous infusion 2,400 mg/m2) will be delivered for 8 weeks (D1=D15).
Other: Early tumor response evaluation by MRI volumetry — Two weeks after the CT completion, the tumor volume will be measured by MRI with specific software which automatically borders the tumor so as to determine the early tumor response. A centralized reassessment of all MRI exams will be systematically performed by two radiologists of the coordinator center.
Radiation: Radiochemotherapy Cap 50 — RCT Cap 50 will combine radiotherapy at a dose of 50 Gy by either conventional 3D or IMRT (2 Gy per fraction, 5 fractions per week during 5 weeks / 44 Gy in mini pelvis, and boost 6 Gy on reduced peritumoral volume) with concomitant oral capecitabine at 1600 mg/m2 per day delivered the days of RT treatment (2 daily intake).
  Arms: Arm B: RCT Cap 50 and then rectal surgery; Arm C: RCT Cap 50 and then rectal surgery
Radiation: Radiochemotherapy Cap 60 — RCT Cap 60 will combine radiotherapy at a dose of 60 Gy by either conventional 3D or IMRT (2 Gy per fraction, 5 fractions per week during 6 weeks / 44 Gy in mini pelvis, and boost 16 Gy on reduced peritumoral volume) with concomitant oral capecitabine at 1600 mg/m2 per day delivered the days of RT treatment (2 daily intake)
  Arms: Bras D: RCT Cap 60 and then rectal surgery
Procedure: Radical proctectomy with total mesorectal excision — The proctectomy can be performed by laparoscopic surgery or conventional laparotomy.

SUMMARY:
The purpose of this study is to determine whether the tailored management of locally advanced rectal carcinoma can improve the oncologic and functional outcome.

DETAILED DESCRIPTION:
Locally advanced rectal carcinoma raise the issue of both the oncological control, local and general, and the therapeutic morbidity. Surgery alone can cure only one out of two patients, radiochemotherapy improves the local control but the metastatic risk remains about 30% with enhanced postoperative morbidity and poor functional results. The tumor response to preoperative treatment is the major prognostic factor which revealed the aggressiveness of the tumor. To this day, there are no biologic predictive markers for tumor response.

The purpose of this trial is to tailor the management according to the early tumoral response after short and intensive induction trichemotherapy. MRI volumetric tumor response will be used to distinguish between good responders and bad responders.

"Very good" responders will be randomized to either immediate surgery or radiochemotherapy followed by surgery (Standard arm: Cap 50). "Good or bad" responders will be randomized between two arms: intensive radiochemotherapy (Cap 60) or the standard arm (Cap 50).

This tailored management should result in a better oncologic prognosis with a lower rate of post therapeutic functional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal carcinoma
* Primary tumor evaluated by pelvic MR Imaging:

  i) iT3 ≥c tumors, with MRI showing a predictive CRM ≤ 2 mm or a EMS (Extra Mural Spread) ≥ 5 mm

ii) Resectable iT4 tumors (only randomized within the "poor responders" group)

iii) Any T tumors with MRI showing a predictive CRM ≤ 1 mm

* No detectable metastases: Thorax-abdomen-pelvic CT-scan
* Patient ≥ 18 years
* ECOG Performance Status 0-1-2
* Patient information and written informed consent form signed
* Patient who can receive radiotherapy and chemotherapy
* Negative pregnancy test in women of childbearing potential
* Patient covered by a Social Security system
* Hematology : Haemoglobin ≥ 9 g/dL, WBC ≥ 4000/mm3, neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Hepatic function : total bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 3 x ULN, Alkaline phosphatases ≤ 3 x ULN
* Renal function : creatinine ≤ 1.25 x ULN or creatinine clearance ≥ 60 ml/min

Exclusion Criteria:

* Indication for immediate surgery
* Primary tumor not measured at the MRI before inclusion
* Previous pelvic radiotherapy
* Contraindication to radiotherapy and/or chemotherapy
* Severe renal or liver impairment
* Cardiac and/or coronary disease which could contraindicate 5-Fu administration
* Active infectious disease
* Peripheral sensitive neuropathy
* History of prior cancer (except if it was cured more than 5 years ago, and if complete remission)
* Patient (male or female) of reproductive potential not using an effective contraceptive method during the whole treatment and up to 6 months after the completion of treatment
* Concurrent participation in any other clinical trial likely to interfere with the therapeutic schedule
* Fertile female patient not using adequate contraception, or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Ro resection rate | Within 15 days after surgery
  To confirm the feasibility of a tailored management with a 90% R0 resection rate achieved for all arms.

SECONDARY OUTCOMES:
Efficiency of MRI for prognosis | Within 15 days after the surgery
  To specify the efficiency of MRI for prognosis in terms of volumetry, downstaging, downsizing and CRM measurement after completion of the induction trichemotherapy.
Compliance rate with neoadjuvant treatment schedule | Within 4 months after the start of treatment
  To measure the compliance rate to the whole neoadjuvant schedule (induction CT + radiochemotherapy)
Acute and late toxicity of neoadjuvant treatments | For the duration of treatment, as expexcted to be up to 4 months and within the 5-year follow-up
  To evaluate overall toxicity of neoadjuvant treatments (induction trichemotherapy + radiochemotherapy) according to the Common Terminology Criteria for Adverse Events v4.0 (NCI CTC v4.0).
Pathological complete response rate | Within 15 days after surgery
  To assess the pathological complete response rate (ypT0N0)
Tumor regression grade (TRG) | Within 15 days after surgery
  To assess at pathologic examination the tumor regression grade (TRG) according to the Dworak classification.
Perioperative and postoperative morbidity | Within 6 weeks after surgery and during the 5-year follow-up
  To assess the impact of the therapeutic strategy on perioperative and postoperative morbidity.
Sphincter-saving surgery rate | Up to 2 months after the end of the neoadjuvant treatment
  To assess the impact of the therapeutic strategy on the rate of sphincter-saving surgery.
Functional outcome | For a 5-year follow-up
  To assess the long-term digestive,urinary and sexual functional results of tailored strategy
Quality of life | For a 5-year follow-up
  To assess the impact of treatments on quality of life according to the EORTC QLQ-C30.
Local recurrence rate | For a 5-year follow-up
  To measure the local recurrence rate in each treatment arm.
Incidence of metastases | For a 5-year follow-up
  To measure the incidence of distant metastases (liver, pulmonary, peritoneal, ganglionnary or any others) in each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUANET, MD, Ph D, Principal Investigator — CRLC Val d'Aurelle-Paul Lamarque
Locations (1):
- CRLC Val d'Aurelle-Paul Lamarque, Montpellier, France

REFERENCES:
- [Derived] Rouanet P, Rullier E, Lelong B, Maingon P, Tuech JJ, Pezet D, Castan F, Nougaret S; GRECCAR Study Group*. Tailored Strategy for Locally Advanced Rectal Carcinoma (GRECCAR 4): Long-term Results From a Multicenter, Randomized, Open-Label, Phase II Trial. Dis Colon Rectum. 2022 Aug 1;65(8):986-995. doi: 10.1097/DCR.0000000000002153. Epub 2022 Jul 5. PMID 34759247
- [Derived] Rouanet P, Rullier E, Lelong B, Maingon P, Tuech JJ, Pezet D, Castan F, Nougaret S; and the GRECCAR Study Group. Tailored Treatment Strategy for Locally Advanced Rectal Carcinoma Based on the Tumor Response to Induction Chemotherapy: Preliminary Results of the French Phase II Multicenter GRECCAR4 Trial. Dis Colon Rectum. 2017 Jul;60(7):653-663. doi: 10.1097/DCR.0000000000000849. PMID 28594714